CLINICAL TRIAL: NCT04876612
Title: Effect of Limaprost in Combination With Transforaminal Epidural Steroid Injection for the Treatment of Lumbar Spinal Stenosis: a Prospective, Double-blind, Randomized Controlled Trial
Brief Title: Effect of Limaprost in Combination With Transforaminal Epidural Steroid Injection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyoun Moon, Associate Professor, Seoul National University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2102-086-119
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients who received placebo after transforminal epidural steroid injection (Placebo Comparator): Patients who took placebo for 12 weeks after TFESI
  Interventions: Procedure: Transforaminal epidural steroid injection (TFESI)
- Patients who received limaprost (Opalmon®) after transforaminal epidural steroid injection (Experimental): Patients who took limaprost (Opalmon®) for 12 weeks after TFESI
  Interventions: Procedure: Transforaminal epidural steroid injection (TFESI)

INTERVENTIONS:
Procedure: Transforaminal epidural steroid injection (TFESI) — Well trained pain physician performs all the fluoroscopy-guided transforaminal epidural steroid injection (TFESI), who is not involved in evaluating study variables. Electrocardiography, noninvasive blood pressure, heart rate, and peripheral oxygen saturation were monitored for all patients before, while, and after conducting procedure. For TFESI, patients are prone positioned, and skin preparation on injection site is done with chlorohexidine. Procedure is conducted under fluoroscopy guidance at the patient's symptom complaining level. After confirming with a contrast medium, 3 ml of 0.1875% ropivacaine and 5 mg of dexamethasone are administered.

SUMMARY:
The purpose of this study was to compare the effects of limaprost(Opalmon® ) on walking ability, low back pain and leg pain after transforaminal epidural steroid injection (TFESI) was administered compared to the placebo group.

DETAILED DESCRIPTION:
This study is a prospective, randomized, comparative clinical study that is assigned to a placebo group or a trial group before transforaminal epidural steroid injection (TFESI) is performed.

The subjects of the study will receive an explanation of the study and decide to participate voluntarily in patients who have decided to undergo TFESI for neurogenic claudication and low back pain or leg pain due to lumbar spinal canal stenosis (LSS).

All study subjects are presented with TFESI at the level appropriate for their symptoms in the operating room and then returned to the recovery room. All participants will be monitored for non-invasive blood pressure, electrocardiography, heart rate, and peripheral oxyven saturation during and after the procedure.

Patients assigned to the placebo group will take placebo three times a day and one tablet once from the first day after receiving TFESI. Patients assigned to the trial group will take limaprost (Opalmon®) three times a day, one tablet once from the first day after receiving TFESI. In both groups, the drug was administered for 12 weeks.

In both groups, during the first 4 weeks, no drug changes or additional procedures were observed, and only Acetaminophen was allowed as a rescue drug.

After TFESI, visits at 4 weeks, 8 weeks and 12 weeks to collect each measurement variable.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 to 85 years

Patients with a new or known diagnosis of lumbar spinal stenosis on Magnetic Resonance Imaging (MRI)

Patients scheduled to undergo TFESI due to low back pain or leg pain

Exclusion Criteria:

Refusal of a patient

Coagulopathy

Systemic infection or local infection at the needle injection site

Patients with lumbar instability

Neoplasms in the needle path

Allergy to amide-type local anesthetics

Decreased cognition to the extent that NRS is incomprehensible

Patients with peripheral vascular disease (including peripheral arterial disease)

Patients taking anticoagulant or antiplatelet drugs

Patients with severe cardiovascular disease or liver or kidney disease

Patinets with cerebral infarction

Patinets with a history of gastrointestinal bleeding

Patinets who have had lumbar spine surgery or are expected to receive it within 12 months

Patients who show positive in the straight leg elevation test

Patients who are allergic or sensitive to limaprost (Opalmon®) and placebo or their ingredients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
ODI (Oswestry Disability Index) change | 4 weeks after placebo or limaprost (Opalmon®)
  The change in ODI compared to the baseline was measured at the outpatient visit.

SECONDARY OUTCOMES:
ODI (Oswestry Disability Index) change | 8 weeks after placebo or limaprost (Opalmon®)
  The change in ODI compared to the baseline was measured at the outpatient visit.
ODI (Oswestry Disability Index) change | 12 weeks after placebo or limaprost (Opalmon®)
  The change in ODI compared to the baseline was measured at the outpatient visit.
Treadmill test change | 4 weeks after placebo or limaprost (Opalmon®)
  The change in treadmill test compared to the baseline was measured at the outpatient visit.
Treadmill test change | 8 weeks after placebo or limaprost (Opalmon®)
  The change in treadmill test compared to the baseline was measured at the outpatient visit.
Treadmill test change | 12 weeks after placebo or limaprost (Opalmon®)
  The change in treadmill test compared to the baseline was measured at the outpatient visit.
Numeric Rating Scale (NRS) change | 4 weeks after placebo or limaprost (Opalmon®)
  The change in NRS compared to the baseline was measured at the outpatient visit.
Numeric Rating Scale (NRS) change | 8 weeks after placebo or limaprost (Opalmon®)
  The change in NRS compared to the baseline was measured at the outpatient visit.
Numeric Rating Scale (NRS) change | 12 weeks after placebo or limaprost (Opalmon®)
  The change in NRS compared to the baseline was measured at the outpatient visit.
Euroqol-5 Dimensions Questionnaire (EQ-5D) change | 4 weeks after placebo or limaprost (Opalmon®)
  The change in EQ-5D compared to the baseline was measured at the outpatient visit.
Euroqol-5 Dimensions Questionnaire (EQ-5D) change | 8 weeks after placebo or limaprost (Opalmon®)
  The change in EQ-5D compared to the baseline was measured at the outpatient visit.
Euroqol-5 Dimensions Questionnaire (EQ-5D) change | 12 weeks after placebo or limaprost (Opalmon®)
  The change in EQ-5D compared to the baseline was measured at the outpatient visit.
Beck Depression Inventory (BPI) change | 4 weeks after placebo or limaprost (Opalmon®)
  The change in BPI compared to the baseline was measured at the outpatient visit.
Beck Depression Inventory (BPI) change | 8 weeks after placebo or limaprost (Opalmon®)
  The change in BPI compared to the baseline was measured at the outpatient visit.
Beck Depression Inventory (BPI) change | 12 weeks after placebo or limaprost (Opalmon®)
  The change in BPI compared to the baseline was measured at the outpatient visit.
Changes in analgesic drugs | 12 weeks after placebo or limaprost (Opalmon®)
  The change in analgesic drugs compared to the baseline was measured at the outpatient visit.

CONTACTS AND LOCATIONS:
Overall Officials: Youn Moon Jee, MD, PhD, Study Director — Seoul National University Hospital; Jeongsoo Kim, MD, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No